CLINICAL TRIAL: NCT03768271
Title: French Cohort on the Becoming of Recent Articular Psoriatic Rheumatism (A Psoriatic Arthritis CoHort)
Brief Title: APACHE Cohort (A Psoriatic Arthritis CoHort)
Acronym: APACHE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180024
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: Cohort Study; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, urine, DNA, RNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoriatic arthritis (PsA) is a chronic inflammatory rheumatic disease, belonging to the wide spectrum of spondyloarthritis, but with the particularity to be associated with personal psoriasis or familial psoriasis. PsA can be a very disabling disease through progressive and irreversible joint damage. Long-term functional prognosis of patients with PsA is correlated with the presence and severity of the radiographic joint lesions of the disease.

However, the proportion of patients who will develop those peripheral joint damages is not yet known and less over the factors which are associated/involved in such an aggressive pattern of the disease. Early identification of this subgroup of patients is particularly important for determining early "intensive" treatment, strict management with a Treat To Target approach, and identification of new treatments with a stronger structural effect.

The main objective of this prospective 10 years cohort is to describe the 5 years structural (radiographic) severity of recent PsA with recent peripheral arthritis.Some of the secondary objectives are to describe the 10 years structural severity within those patients, and to determine the predictive factors of those 5 and 10 years radiographic lesions (genetic, environmental, clinic, therapeutic factors).

APACHE will provide a unique longitudinal standardized database concerning patients with PsA with very recent peripheral arthritis. Research projects which will based on those collected data should allow to identify the mechanisms of aggressive joint damage, to highlight mew treatments targets, to better describe the burden of the disease, to test previous or develop new assessments tolls, to develop early diagnostic criteria

DETAILED DESCRIPTION:
Method:APACHE is a prospective national multicentre (29) cohort including and following during 10 years patients with a first peripheral arthritis in the past year, attributing to a PsA according to the treating rheumatologist. 425 patients will be included during a 4 years period before the follow-up. Standardized visits are planned throughout the 10 years follow-up, permitting the collection of various data:

* clinical data
* Patients Reported Outcome
* usual lab parameters
* plasma, serum and urines
* Baseline and one year RNA, DNA
* peripheral X-Rays, Ultrasounds and MRI at different time points Those visits have non interventional character (no therapeutic decision will be taken) Those collected data will allow submissions of many research projects to the scientific committee of the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Women or men aged from 18 to 60 inclusive
* First episode of peripheral arthritis in the last 12 months, authenticated by a rheumatologist
* Psoriasis diagnosed by a practitioner or family history of psoriatic arthritis (first-degree relative [parent or sibling] or second degree relative)
* Arthritis most likely recognized as a psoriatic arthritis by a rheumatologist (diagnostic confidence score : ≥ 7 out of 10)
* Signed informed consent form
* Affiliation to a social security system

Exclusion Criteria:

* Formal diagnostic of inflammatory rheumatism other than psoriatic arthritis
* Treatment or history of treatment with a biomedicine
* Patient receiving csDMARDS or apremilast treatment for 1 year or more
* Patient having received csDMARDS or apremilast treatment during the last 12 months
* Oral steroids in the last 4 weeks, above 10 mg/d of prednisone or with modified dosage
* intravenous or intra articular steroids in the last 4 weeks
* IRM contraindication
* Cognitive, mental or psychic disorders impeding protocol accomplishment
* Difficulties with French language understanding
* Patient under tutorship or curatorship
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with peripheral psoriatic arthritis diagnosed at an early stage.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at least one erosion on the 5-years X-Rays | at 5 years
  The primary endpoint is the presence / absence of at least one erosion on at least one of the 5-years X-Rays, i.e., wrists and hands, feet, and if present other joint(s) with arthritis at baseline.
  The assessment of erosions will be done by 3 trained readers.

SECONDARY OUTCOMES:
Percentage of patients with at least one joint space narrowing and one periostitic lesion on the 5-years X-Rays. | at 5 years
  this endpoint is the presence of at least one joint space narrowing and one periostitic lesion on at least one of the 5-years X-Rays, i.e., wrists and hands, feet, and if present other joint(s) with arthritis at baseline. The assessment of erosions will be done by 3 trained readers.
Percentage of patients with at least one erosion, joint space narrowing, periostitic lesion, on the 10-years X-Rays. | at 10 years
  this endpoint is the presence of at least one erosion, joint space narrowing, periostitic lesion, on at least one of the 10-years X-Rays, i.e., wrists and hands, feet, and if present other joint(s) with arthritis at baseline. The assessment of erosions will be done by 3 trained readers.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle VIVALDO, Study Chair — DRCD-Assistance Publique des Hôpitaux de Paris
Locations (3):
- France (3):
  - Henri-Mondor Hospital, Créteil
  - Lapeyronie Hospital, Montpellier
  - Saint Joseph Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claudepierre P, Gaujoux-Viala C, Constantin A, Berenbaum F, Combe B, Devauchelle V, Goupille P, Richette P, Wendling D, Mouterde G, Pascart T, Razat B, Audureau E, Jousse-Joulin S, Gossec L. Early peripheral psoriatic arthritis: Baseline features of the first 186 patients in the French Nationwide APACHE Cohort. Joint Bone Spine. 2025 Dec;92(6):105930. doi: 10.1016/j.jbspin.2025.105930. Epub 2025 May 27. PMID 40441347